CLINICAL TRIAL: NCT02195349
Title: A Randomised, Double Blind (Sponsor Unblinded), Placebo-controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a IV Dose of GSK2831781 in Healthy Volunteers and Patients With Plaque Psoriasis
Brief Title: A First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Intravenous (IV) Dose of GSK2831781 in Healthy Volunteers and Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200630; 2014-000312-33 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: Tuberculin Purified Protein Derivative; Delayed Type Hypersensitivity; Biopsy; Induration; First time in human; T-cells; LAG-3; safety; GSK2831781; psoriasis
MeSH Terms: conditions — Psoriasis; Hypersensitivity, Delayed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Subjects (no DTH) (Experimental): One subject will be dosed with GSK2831781 (0.0003 mg/kg) and one with placebo. Depending on the safety data obtained for 28 days post dose along with the available PK data, a dose escalation may be done to the next planned dose (0.0015 , 0.0075, 0.04, 0.15 mg/kg). In case safety findings are noted then the cohort may be expanded to a maximum cohort size of 6:3 (GSK2831781: placebo) or the escalation will be stopped.
  Interventions: Biological: GSK2831781; Biological: Placebo
- Healthy Subjects (DTH) (Experimental): Sentinel subjects (one dosed with GSK2831781 (0.0003 mg/kg) and one with placebo) will be used in the cohort. Following a review of safety data up to 48 hours post dose, an additional 5 active (GSK2831781) and 1 placebo subject will be dosed (no more than 2 subjects per day with dosing separated by at least 1 hour). After reviewing the safety data for 28 days the healthy subjects (DTH) will be escalated to the planned dose of GSK2831781 (0.0075, 0.04, 0.15 mg/kg) in 6:3 ratio with placebo.
  Interventions: Biological: GSK2831781; Biological: Placebo
- Subjects with Psoriasis (Experimental): Sentinel subjects (one dosed with GSK2831781 and one with placebo) will be used in the cohort. Following a review of safety data up to 48 hours post dose, an additional 5 active (GSK2831781) and 2 placebo subjects will be dosed (no more than 2 subjects per day with dosing separated by at least 1 hour). All subsequent cohorts do not require stratification for pre-existing ADAs. After reviewing the safety data for 28 days for minimum of 8 out of 9 subjects within the cohort and all subjects have completed dosing and the inpatient monitoring until Day 4, the subjects with psoriasis will be escalated to the planned dose of GSK2831781 (1.5 and 5 mg/kg) in 6:3 ratio with placebo.
  Interventions: Biological: GSK2831781; Biological: Placebo

INTERVENTIONS:
Biological: GSK2831781 — GSK2831781 (100 milligram (mg)/mL) and its dilutions (Diluent - 0.9 percent saline solution containing 0.015 percent Polysorbate 80) as clear or opalescent, colourless, yellow to brown liquid solution administered by IV over approximately 2 hours.
Biological: Placebo — Commercial saline solution administered by IV over approximately 2 hours

SUMMARY:
This study is a phase I, randomised, double blind (sponsor unblinded), placebo-controlled, single ascending dose study GSK2831781 administered by IV. GSK2831781 is a humanized Antibody Dependent Cell Cytotoxicity (ADCC) enhanced monoclonal afucosylated antibody that is specific to the Lymphocyte Activation Gene-3 (LAG-3) protein. This is the first administration of GSK2831781 in humans and will evaluate in two parts the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of single IV doses of GSK2831781 administered to healthy subjects previously vaccinated with Bacillus Calmette Guérin (BCG) (Part A delayed type hypersensitivity [DTH] cohorts) and patients with plaque psoriasis (Part B). The inclusion of DTH and psoriasis subjects to explore the mechanism in biopsies and clinical response endpoints in these populations, as well as investigate systemic biomarkers will provide useful information prior to conducting studies in other immune-inflammatory disease which will involve more invasive tissue biopsies. Measuring the pharmacology of GSK2831781 using the depletion of LAG-3+ T-cells in skin biopsies from Tuberculin Purified Protein Derivative (PPD) skin challenge and lesional skin biopsies from patients with psoriasis, will be helpful in understanding of the dose response relationship, which will be important for designing future studies in immuno-inflammatory diseases, including psoriasis. Approximately 67 subjects will be enrolled to complete dosing and critical assessments. The subject numbers will be split to approximately 40 healthy subjects (Part A) and 27 patients with psoriasis (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Part A males aged between 18 and 65 years of age and Part B males and females aged between 18 and 75 years of age inclusive, at the time of signing the informed consent
* Part A: A body weight <=120 kilogram (kg) and Body mass index (BMI) within the range 19-32 kg/square meter (m^2) (inclusive), Part B: BMI within range 19-35 kg/m^2 (inclusive).
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent)
* Based on single or averaged Electrocardiogram QT interval corrected for heart rate (QTc) values of triplicate Electrocardiogram (ECGs) obtained over a brief recording period: Electrocardiogram QT interval corrected for heart rate using Fridericia's formula (QTcF) <450 milliseconds (msec)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

For Part A study subjects only

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECGs. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the Glaxosmithkline (GSK) Medical Monitor, if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures

Delayed type hypersensitivity (DTH) cohorts only

* Subjects with a history of Bacillus Calmette Guérin (BCG) vaccination as evidence by either: A BCG scar and verbal confirmation of BCG vaccination ; Or documented medical history of a BCG vaccination with or without a BCG scar
* Subjects with a history of current vaccination for Tetanus, diphtheria, measles, pertussis, mumps and rubella

For Part B study subjects only

* Subject has psoriasis covering Body Surface Area (BSA) >=3 percent as assessed at Screening and Day-1
* Subject has had a confirmed diagnosis of chronic plaque-type psoriasis (without recent documented flare within 30 days prior to screening) for at least 6 months
* Subject has at least 2 stable plaques assessed at Screening and Day -1. One of a suitable size and in a site suitable for repeat biopsy, and one for index lesion Plaque Lesional Severity Score (PLSS) scoring. Both must have a PLSS lesional score of >=2 for the induration component (moderate or above), >=1 for erythema and scaling with a total score of >=5. The biopsy lesion must not be on the face, groin or scalp and must be protected from the sun
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screening and negative urine hCG test at Day -1 for Females of Reproductive Potential [FRP]), not lactating, and at least one of the given conditions applies: Non-reproductive potential defined as pre-menopausal females with a documented tubal ligation; or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; or hysterectomy; or documented bilateral oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to use a barrier method (male condom or female diaphragm) plus to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP from 28 days prior to the first dose of study medication and until completion of the follow-up visit.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. The investigator or designee should remind the subjects of the need to comply with these requirements approximately monthly, either at study visits or by telephone call until the follow-up visit.

Exclusion Criteria:

* Received live vaccine (s) attenuated or recombinant within 4 weeks of Day 1 or plan to receive a live vaccination during the study until follow-up
* Subjects from a high risk area of the world for tuberculosis or have history of tuberculosis or have close family members with confirmed Mycobacterium tuberculosis (MTB) infection or positive at screening by Quantiferon testing
* Subject is unable to abstain from travelling to areas with high endemic rates of infectious diseases until the end of the follow up period
* A medical history of severe allergic reaction, angio-edema, anaphylaxis or immunodeficiency
* Subjects with neutrophil results below the normal range at screening and baseline
* Subjects with any clinical, even mild, Gastrointestinal (GI) upset such as, but not limited to, diarrhea or abdominal cramping during the previous week before dosing, as well as history of more chronic GI upset, e.g. Irritable Bowel Syndrome (IBS)
* Current evidence of ongoing or acute infection within 3 months prior to the first dose of study drug, such as: Serious local infection (e.g. cellulitis, abscess); Systemic infection [e.g. pneumonia, septicaemia, Tuberculosis (TB)]
* Subjects who test positive for pre-existing ADA to GSK2831781 at screening.
* History of malignancy, except for basal cell or squamous cell carcinoma, or in situ cervical carcinoma that has been fully treated and shows no evidence of recurrence
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8gram (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* History of sensitivity to any of the study medications or Tuberculin Purified Protein Derivative (PPD) challenge agent, or components thereof or a history of drug (or Immunoglobulin G therapeutic antibodies) or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen
* A positive test for Human Immunodeficiency Virus (HIV) antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Subjects with an aspartate aminotransferase and/or gamma glutamyltransferase level above the upper limit of normal at screening and/or baseline will be excluded

For Part A study subjects only

* Use of prescription drugs or non-prescription drugs, if in the opinion of the investigator (in consultation with the GSK medical monitor), the medication will interfere with the study procedures or compromise subject safety
* Subjects must not currently be taking any of the following: topical steroids on the arms, oral or systemic steroids or any other immune-modulators (the washout period will be determined, on a case by case basis, by the investigator in consultation with the GSK medical monitor)
* Subjects with an aspartate aminotransferase and/or gamma glutamyltransferase level above the upper limit of normal at screening and/or baseline will be excluded.

For Part A (only cohorts with DTH challenge) study subjects only:

* Use of nicotine patches on the arm at screening that would interfere with the injection sites
* Presence of tattoos, naevi or other skin abnormalities such as keloids (or a history of keloids) that may, in the opinion of the investigator, interfere with DTH assessments
* Subjects participating, within seven days of screening, in recreational sun-bathing, or the use of a sun-bed, on the area of the skin from the wrist to the shoulder (inclusive)

For Part B study subjects only:

* History of significant cardiac, endocrinologic, haematologic, pulmonary, metabolic, renal, hepatic, immunologic (excluding psoriasis and psoriatic arthritis), urologic, neurologic, dermatologic (except psoriasis), psychiatric or gastrointestinal conditions that, in the opinion of the investigator and/or GSK medical monitor, places the subject at unacceptable risk
* Clinically significant abnormalities of laboratory assessments (not related to disease) as judged by the investigator and/or GSK medical monitor
* All systemic psoriasis medications, including psoralen long-wave ultraviolet radiation treatments, or other systemic immunosuppressives, are not allowed within 5 half lives prior to Day-1 (Methotrexate and cyclosporin are not allowed within 8 weeks of Day -1; Psoralen long-wave Ultraviolet (UV) is not allowed within 4 weeks of Day-1). Subjects should not be included if the investigator considers that the subject is at high risk of requiring rescue with prohibited medication for duration of study up to follow-up. This assessment should be based on current disease activity or a history of frequent and/or severe flares requiring systemic immunosuppression.
* The use of single treatment phototherapy (ultraviolet B or self treatment with tanning beds) is not allowed within 14 days prior to Day -1
* The use of topical therapies for psoriasis are not allowed with 7 days prior to Day-1 on the index lesion or biopsy plaque
* Previous treatment with anti- Tumour necrosis factor (TNF)/ Interleukin (IL)-12/IL-23 or any other monoclonal antibodies is not allowed within 12 weeks prior to Day-1
* Patients that require narrow therapeutic index medications from Screening to Follow-up
* Vulnerable subjects (e.g. person kept in detention)
* Subjects who are not able to understand and communicate in the native language of the country where the study is conducted.
* Subjects who work for the Sponsor or CRO.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (2):
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20763

REFERENCES:
- [Background] Ellis J, J B Marks D, Srinivasan N, Barrett C, Hopkins TG, Richards A, Fuhr R, Albayaty M, Coenen M, Liefaard L, Leavens K, Nevin KL, Tang S, Hughes SA, Fortunato L, Edwards K, Cui Y, Anselm R, Delves CJ, Charles E, Feeney M, Webb TM, Brett SJ, Schmidt TS, Stone J, Savage COS, Wisniacki N, Tarzi RM. Depletion of LAG-3+ T Cells Translated to Pharmacology and Improvement in Psoriasis Disease Activity: A Phase I Randomized Study of mAb GSK2831781. Clin Pharmacol Ther. 2021 May;109(5):1293-1303. doi: 10.1002/cpt.2091. Epub 2020 Nov 24. PMID 33113155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single ascending dose study conducted in healthy volunteers and participants with plaque psoriasis. Participants were enrolled in Germany and the United Kingdom from 30 July 2014 to 07 March 2018.
Pre-assignment Details: A total of 330 participants were screened in healthy volunteer cohorts and 197 participants in psoriasis cohorts of which 290 were screen failures in healthy volunteer cohorts and 170 in psoriasis cohorts. A total of 40 participants were enrolled in healthy cohorts and 27 in psoriasis cohorts.
Groups:
- Placebo for Healthy Volunteer Combined: Healthy volunteers with no delayed type hypersensitivity (DTH) and with DTH received a single dose of placebo-matching saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.0003 mg/kg (ADA-ve): Healthy volunteers with no DTH and without pre-existing anti-drug antibodies negative (ADA-ve) status received a single dose of GSK2831781 0.0003 milligram per kilogram (mg/kg) saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.0015 mg/kg (ADA-ve): Healthy volunteers with no DTH and without pre-existing ADA-ve status received a single dose of GSK2831781 0.0015 mg/kg saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.0075 mg/kg (ADA-ve): Healthy volunteers with no DTH and without pre-existing ADA-ve status received a single dose of GSK2831781 0.0075 mg/kg saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.04 mg/kg (ADA-ve): Healthy volunteers with no DTH and without pre-existing ADA-ve status received a single dose of GSK2831781 0.04 mg/kg saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.15 mg/kg (ADA-ve): Healthy volunteers received a skin challenge of 0.1 milliliter (mL) of 2 tuberculin unit (TU) or 10 TU purified protein derivative (PPD) (0.04 microgram [mcg]/0.1mL), injected intradermally into the volar aspect of the left and right forearm, once in each forearm on Day 1; followed by a single dose of GSK2831781 0.15 mg/kg saline solution, intravenously on Day 29 for 2 hours post-infusion start in healthy volunteers with DTH and with pre-existing ADA-ve status; further followed by 0.1 mL of 2 TU or 10 TU PPD was injected intradermally into the volar aspect of the left and right forearm, twice in each forearm on Day 29.
- GSK2831781 0.15 mg/kg (ADA+ve): Healthy volunteers with no DTH and without pre-existing ADA+ve status received a single dose of GSK2831781 0.15 mg/kg saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- Placebo for Psoriasis: Psoriasis participants received a single dose of placebo-matching saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.5 mg/kg: Psoriasis participants with pre-existing ADA-ve and ADA+ve status received a single dose of GSK2831781 0.5 mg/kg saline solution, intravenously, on Day 1 for 2 hours post-infusion start.
- GSK2831781 1.5 mg/kg: Psoriasis participants with pre-existing ADA-ve and ADA+ve status received a single dose of GSK2831781 1.5 mg/kg saline solution, intravenously, on Day 1 for 2 hours post-infusion start.
- GSK2831781 5 mg/kg: Psoriasis participants with pre-existing ADA-ve and ADA+ve status received a single dose of GSK2831781 5 mg/kg saline solution, intravenously, on Day 1 for 2 hours post-infusion start.
Period: Overall Study
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Started | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Completed | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo for Healthy Volunteer Combined: Healthy volunteers with no DTH and with DTH received a single dose of placebo-matching saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.0003 mg/kg (ADA-ve): Healthy volunteers with no DTH and without pre-existing ADA-ve status received a single dose of GSK2831781 0.0003 mg/kg saline solution, intravenously on Day 1 for 2 hours post-infusion start.
- GSK2831781 0.15 mg/kg (ADA-ve): Healthy volunteers received a skin challenge of 0.1 mL of 2 TU or 10 TU PPD (0.04 mcg/0.1mL), injected intradermally into the volar aspect of the left and right forearm, once in each forearm on Day 1; followed by a single dose of GSK2831781 0.15 mg/kg saline solution, intravenously on Day 29 for 2 hours post-infusion start in healthy volunteers with DTH and with pre-existing ADA-ve status; further followed by 0.1 mL of 2 TU or 10 TU PPD was injected intradermally into the volar aspect of the left and right forearm, twice in each forearm on Day 29.
- Total: Total of all reporting groups
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg | Total
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 6
  Male | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 5 | 6 | 5 | 5 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 6
  White - White/Caucasian/European heritage | 12 | 1 | 1 | 5 | 5 | 4 | 6 | 9 | 6 | 6 | 6 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance (PCI)
Description: Hematology parameters with PCI ranges: hematocrit (high: >0.54 percentage of red blood cells), hemoglobin (high: >180 grams per liter [g/L]), lymphocytes (low: <0.8*giga cells per liter [10^9/L]), neutrophil count (low: <1.5*10^9/L), platelet count (low: <100*10^9/L and high: >550*10^9/L), and while blood cell count (low: <3*10^9/L and high: >20*10^9/L) for healthy volunteers and psoriasis participants. Safety population consisted of all randomized participants who received at least one dose of study treatment. Only those participants for which at least one value of PCI was reported are summarized.
Time Frame: Up to 307 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of PCI
Description: Clinical chemistry parameters and their potential clinical concern values: albumin (low: <30 millimoles per liter [mmol/L]), calcium (low: <2 mmol/L, high: >2.75 mmol/L), creatinine (high: >44.2 mmol/L), glucose (low: <3 mmol/L, high: >9 mmol/L), magnesium (low: <0.5 mmol/L, high: >1.23 mmol/L), phosphorus (low: <0.8 mmol/L, high: >1.6 mmol/L), potassium (low: <3 mmol/L, high: >5.5 mmol/L), sodium (low: <130 mmol/L, high: >150 mmol/L), and total carbon dioxide (CO2) (low: <18 mmol/L, high: >32 mmol/L). Number of participants with clinical chemistry of PCI are presented.
Time Frame: Up to 307 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 3

3. Primary Outcome: Number of Participants With Vital Signs of PCI
Description: Vital signs included heart rate, systolic and diastolic blood pressure and body temperature were performed with the participant in a semi-supine position after the participant had rested for at least 5 minutes. The PCI range for heart rate (low: <40 beats per minute [BPM] and high: >110 BPM), systolic blood pressure (low: <85 and high: >160 millimeter of mercury [mmHg]), diastolic blood pressure (low: <45 mmHg and high: >100 mmHg) and body temperature (low: <35 degree Celsius and high: >37.5 degree Celsius). Number of participants with vital signs of PCI are presented.
Time Frame: Up to 307 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2

4. Primary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) of PCI
Description: Triplicate ECG was measured in a semi-supine position after 5 minutes rest. A single 12-lead ECG was obtained by using an ECG machine that automatically calculates heart rate and measured PR, QRS, QT, and Fridericia's formula (QTcF) intervals. The PCI ranges for QTc Interval (high: >450 millisecond [msec]), PR Interval (low: <110 msec and high: >220 msec) and QRS Interval (low: <75 msec and high: >110 msec). Number of participants with ECG values of PCI are presented.
Time Frame: Up to 307 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 1

5. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect and other important medical events judged by the investigator that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: Up to 307 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Participants
  Any AEs | 8 | 0 | 0 | 5 | 6 | 3 | 3 | 9 | 4 | 6 | 6
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Change From Baseline in Interleukin (IL)-6, IL-8, Interferon-gamma, and Tumor Necrosis Factor (TNF) Alpha
Description: IL-6, IL-8, interferon-gamma and TNF alpha were assessed at indicated time points. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day 1, pre-dose). Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline, 6, 12, 24 and 48 hours post-dose
Population: Safety population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 14 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
Picogram per milliliter (pg/mL)
  IL-6: 6 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 2.889 (5.5511) | 1.430 (NA) — Standard deviation could not be calculated for one participant. | 0.000 (NA) — Standard deviation could not be calculated for one participant. | 0.258 (1.8234) | 1.025 (1.6945) | 4.305 (5.0046) | 1.142 (1.9865) | 15.003 (29.0749) | 1.445 (1.9297) | 2.062 (1.5145) | 3.837 (6.7895)
  IL-6: 12 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 3.748 (5.0647) | 7.140 (NA) — Standard deviation could not be calculated for one participant. | 0.000 (NA) — Standard deviation could not be calculated for one participant. | 0.127 (3.2387) | 6.408 (11.0052) | 12.302 (10.2985) | 34.603 (42.6294) | 21.447 (26.3310) | 18.943 (26.2127) | 3.150 (2.0492) | 11.893 (16.0968)
  IL-6: 24 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 0.727 (1.5514) | 1.720 (NA) — Standard deviation could not be calculated for one participant. | 0.000 (NA) — Standard deviation could not be calculated for one participant. | -1.272 (3.1149) | 0.522 (1.2778) | 16.748 (28.4330) | 2.710 (5.1169) | 4.284 (9.7552) | 5.825 (9.9881) | 2.737 (1.8897) | 1.987 (5.9878)
  IL-6: 48 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 1.887 (4.1642) | 7.630 (NA) — Standard deviation could not be calculated for one participant. | 0.000 (NA) — Standard deviation could not be calculated for one participant. | -1.493 (3.6579) | 0.000 (0.0000) | 2.193 (3.8186) | -0.657 (1.1306) | -1.091 (1.6867) | -0.460 (1.8092) | 0.163 (0.6664) | -1.145 (2.8564)
  IL-8: 6 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 1.284 (2.7802) | -0.100 (NA) — Standard deviation could not be calculated for one participant. | -0.210 (NA) — Standard deviation could not be calculated for one participant. | 4.302 (2.7723) | 1.752 (3.0055) | 3.657 (4.9829) | 1.847 (2.1026) | 1.518 (3.5960) | 1.522 (2.6497) | 3.157 (3.7276) | 4.063 (3.7411)
  IL-8: 12 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 4.344 (5.4602) | 1.800 (NA) — Standard deviation could not be calculated for one participant. | 2.760 (NA) — Standard deviation could not be calculated for one participant. | 5.487 (5.5182) | 5.107 (3.1582) | 15.155 (21.9139) | 8.110 (10.8187) | 21.774 (55.5319) | 7.425 (13.5089) | 10.667 (6.9406) | 11.120 (6.7124)
  IL-8: 24 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 6.402 (21.1483) | 2.100 (NA) — Standard deviation could not be calculated for one participant. | -0.260 (NA) — Standard deviation could not be calculated for one participant. | 0.560 (2.2738) | 4.780 (10.3055) | 39.248 (50.1491) | 1.710 (1.9256) | 3.321 (8.3425) | 5.993 (14.0442) | 18.330 (22.5892) | 9.208 (13.2078)
  IL-8: 48 hours (n=14,1,1,6,6,6,6,9,6,6,6) | 1.337 (9.4965) | 47.900 (NA) — Standard deviation could not be calculated for one participant. | -0.740 (NA) — Standard deviation could not be calculated for one participant. | 0.028 (0.0694) | -0.212 (2.1383) | -0.425 (2.7328) | 0.382 (1.0779) | -1.901 (1.8197) | -1.140 (2.4624) | 1.047 (2.7193) | 0.300 (3.0864)
  Interferon-gamma:6hours(n=14, 1,1,6,6,6,6,9,6,6,6) | 0.00 (0.000) | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Interferon-gamma:12hours(n=13,1,1,6,6,6,6,9,6,6,6): number analyzed (Participants) | 13 | 1 | 1 | 6 | 6 | 6 | 6 | 9 | 6 | 6 | 6
  Interferon-gamma:12hours(n=13,1,1,6,6,6,6,9,6,6,6) | 0.00 (0.000) | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Interferon-gamma:24hours(n=14,1,1,6,6,6,6,9,6,6,6) | 0.00 (0.000) | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Interferon-gamma:48hours(n=12,1,1,6,6,6,5,9,6,6,6): number analyzed (Participants) | 12 | 1 | 1 | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6
  Interferon-gamma:48hours(n=12,1,1,6,6,6,5,9,6,6,6) | 0.00 (0.000) | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (NA) — Standard deviation could not be calculated for one participant. | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  TNF alpha:6hours (n=14,1,1,6,6,6,6,9,6,6,6) | 0.166 (1.1347) | 0.050 (NA) — Standard deviation could not be calculated for one participant. | 1.940 (NA) — Standard deviation could not be calculated for one participant. | 4.958 (3.8080) | 3.047 (5.0083) | 5.162 (4.6045) | 1.512 (1.3042) | -0.402 (1.4406) | 2.658 (1.7619) | 2.678 (1.6019) | 3.455 (1.7634)
  TNF alpha: 12 hours (n=14,1,1,6,6,6,6,9,6,6,6) | -0.201 (1.3961) | -1.030 (NA) — Standard deviation could not be calculated for one participant. | 0.700 (NA) — Standard deviation could not be calculated for one participant. | 5.075 (2.8043) | 6.735 (3.9483) | 6.768 (5.9501) | 2.272 (1.5898) | -0.301 (0.5766) | 2.100 (1.9397) | 4.265 (2.6663) | 2.753 (1.1083)
  TNF alpha: 24 hours (n=14,1,1,6,6,6,6,9,6,6,6) | -0.244 (1.4101) | -0.450 (NA) — Standard deviation could not be calculated for one participant. | 0.310 (NA) — Standard deviation could not be calculated for one participant. | 2.650 (1.2128) | 5.935 (3.4483) | 5.372 (4.2010) | 0.883 (2.1105) | -0.029 (1.0534) | 2.775 (1.2677) | 2.942 (2.4473) | 2.502 (1.7958)
  TNF alpha: 48 hours (n=14,1,1,6,6,6,6,9,6,6,6) | -0.366 (1.2390) | 0.420 (NA) — Standard deviation could not be calculated for one participant. | -0.480 (NA) — Standard deviation could not be calculated for one participant. | 0.810 (1.5676) | 0.878 (0.8027) | 1.825 (1.5788) | -0.007 (1.7897) | 0.286 (1.1455) | 0.752 (0.9434) | 1.712 (1.1398) | 1.083 (0.8472)

7. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick in Placebo Healthy Volunteers
Description: Urine samples were collected at indicated time points to analyze parameters including glucose, protein, blood, leucocytes, nitrites and ketones by dipstick. Urine dipstick tests were either read as qualitative concentrations as Negative, Trace, 1+ (low concentrations present), 2+ (moderate concentrations present), 3+ (high concentrations present) and 4+ (very high concentrations present); or as semi quantitative cell counts or concentrations (0, 0.25, 0.5, 1.5,5, 7, 9, 10, 25, 50, 150, 250) where units depend on the test performed; (cells/micro liter for blood and leucocytes; mmol/L for glucose and ketones; g/L for protein), and Negative (not detected) or Positive (detected) for nitrites. For each methodology, abnormal results were defined as those that were not 'Negative' or 'Trace'. Only categories with abnormal urinalysis values are presented.
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 191
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined
Number analyzed (Participants) | 14
Participants
  Occult blood: 6 hours, 0 | 2
  Occult blood: 6 hours, 1+ | 2
  Occult blood: 6 hours, 10 | 1
  Occult blood: 6 hours, 7 | 1
  Occult blood: 12 hours, 0 | 4
  Occult blood: 12 hours, 2+ | 1
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 2
  Occult blood: 72 hours, 1+ | 1
  Occult blood: 72 hours, 10 | 2
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 4
  Occult blood: 168 hours, 1+ | 1
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 4
  Occult blood: Day 22, 0: number analyzed (Participants) | 12
  Occult blood: Day 22, 0 | 4
  Occult blood: Day 22, 10: number analyzed (Participants) | 12
  Occult blood: Day 22, 10 | 0
  Occult blood: Day 22, 2+: number analyzed (Participants) | 12
  Occult blood: Day 22, 2+ | 1
  Occult blood: Day 29, 0: number analyzed (Participants) | 13
  Occult blood: Day 29, 0 | 4
  Occult blood: Day 29, 1+: number analyzed (Participants) | 13
  Occult blood: Day 29, 1+ | 1
  Occult blood: Day 29, 10: number analyzed (Participants) | 13
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 2+: number analyzed (Participants) | 13
  Occult blood: Day 29, 2+ | 1
  Occult blood: Day 29, 25: number analyzed (Participants) | 13
  Occult blood: Day 29, 25 | 0
  Occult blood: Day 43, 0: number analyzed (Participants) | 12
  Occult blood: Day 43, 0 | 4
  Occult blood: Day 43, 1+: number analyzed (Participants) | 12
  Occult blood: Day 43, 1+ | 1
  Occult blood: Day 43, 10: number analyzed (Participants) | 12
  Occult blood: Day 43, 10 | 0
  Occult blood: Day 43, 25: number analyzed (Participants) | 12
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 57, 0: number analyzed (Participants) | 12
  Occult blood: Day 57, 0 | 4
  Occult blood: Day 57, 1+: number analyzed (Participants) | 12
  Occult blood: Day 57, 1+ | 1
  Occult blood: Day 57, 10: number analyzed (Participants) | 12
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 85, 0: number analyzed (Participants) | 10
  Occult blood: Day 85, 0 | 4
  Occult blood: Day 85, 10: number analyzed (Participants) | 10
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 121, 0: number analyzed (Participants) | 10
  Occult blood: Day 121, 0 | 4
  Occult blood: Day 121, 1+: number analyzed (Participants) | 10
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10: number analyzed (Participants) | 10
  Occult blood: Day 121, 10 | 0
  Occult blood: Day 191, 0 | 4
  Occult blood: Day 191, 10 | 0
  Occult blood: Day 191, 25 | 0
  Glucose: 6 hours, 0 | 2
  Glucose: 6 hours, 17 | 1
  Glucose: 6 hours, 7 | 1
  Glucose: 12 hours, 0 | 4
  Glucose: 72 hours, 0 | 3
  Glucose: 72 hours, 3 | 1
  Glucose: 168 hours, 0 | 4
  Glucose: Day 15, 0 | 4
  Glucose: Day 22, 0: number analyzed (Participants) | 12
  Glucose: Day 22, 0 | 4
  Glucose: Day 29, 0: number analyzed (Participants) | 13
  Glucose: Day 29, 0 | 4
  Glucose: Day 43, 0: number analyzed (Participants) | 12
  Glucose: Day 43, 0 | 4
  Glucose: Day 57, 0: number analyzed (Participants) | 12
  Glucose: Day 57, 0 | 4
  Glucose: Day 85, 0: number analyzed (Participants) | 10
  Glucose: Day 85, 0 | 4
  Glucose: Day 121, 0: number analyzed (Participants) | 10
  Glucose: Day 121, 0 | 4
  Glucose: Day 191, 0 | 4
  Ketones: 6 hours, 0 | 3
  Ketones: 6 hours, 7 | 1
  Ketones: 12 hours, 0 | 4
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 4
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 4
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 1
  Ketones: Day 15, 0 | 3
  Ketones: Day 15, 0.5 | 1
  Ketones: Day 22, 0: number analyzed (Participants) | 12
  Ketones: Day 22, 0 | 3
  Ketones: Day 22, 0.5: number analyzed (Participants) | 12
  Ketones: Day 22, 0.5 | 1
  Ketones: Day 29, 0: number analyzed (Participants) | 13
  Ketones: Day 29, 0 | 4
  Ketones: Day 29, 0.5: number analyzed (Participants) | 13
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 43, 0: number analyzed (Participants) | 12
  Ketones: Day 43, 0 | 4
  Ketones: Day 43, 0.5: number analyzed (Participants) | 12
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1.5: number analyzed (Participants) | 12
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0: number analyzed (Participants) | 12
  Ketones: Day 57, 0 | 4
  Ketones: Day 85, 0: number analyzed (Participants) | 10
  Ketones: Day 85, 0 | 3
  Ketones: Day 85, 0.5: number analyzed (Participants) | 10
  Ketones: Day 85, 0.5 | 1
  Ketones: Day 121, 0: number analyzed (Participants) | 10
  Ketones: Day 121, 0 | 4
  Ketones: Day 121, 0.5: number analyzed (Participants) | 10
  Ketones: Day 121, 0.5 | 0
  Ketones: Day 121, 2+: number analyzed (Participants) | 10
  Ketones: Day 121, 2+ | 1
  Ketones: Day 191, 0 | 4
  Ketones: Day 191, 0.5 | 0
  Ketones: Day 191, 1+ | 0
  Nitrite: Day 15, positive | 1
  Nitrite: Day 85, positive: number analyzed (Participants) | 10
  Nitrite: Day 85, positive | 1
  Nitrite: Day 121, positive: number analyzed (Participants) | 10
  Nitrite: Day 121, positive | 1
  Protein: 6 hours, 0 | 3
  Protein: 6 hours, 7 | 1
  Protein: 12 hours, 0 | 4
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 4
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 4
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 1
  Protein: Day 15, 0 | 4
  Protein: Day 15, 1+ | 1
  Protein: Day 22, 0: number analyzed (Participants) | 12
  Protein: Day 22, 0 | 4
  Protein: Day 22, 1+: number analyzed (Participants) | 12
  Protein: Day 22, 1+ | 1
  Protein: Day 29, 0: number analyzed (Participants) | 13
  Protein: Day 29, 0 | 4
  Protein: Day 29, 1+: number analyzed (Participants) | 13
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0: number analyzed (Participants) | 12
  Protein: Day 43, 0 | 4
  Protein: Day 43, 1+: number analyzed (Participants) | 12
  Protein: Day 43, 1+ | 1
  Protein: Day 57, 0: number analyzed (Participants) | 12
  Protein: Day 57, 0 | 4
  Protein: Day 57, 1+: number analyzed (Participants) | 12
  Protein: Day 57, 1+ | 1
  Protein: Day 85, 0: number analyzed (Participants) | 10
  Protein: Day 85, 0 | 4
  Protein: Day 85, 1+: number analyzed (Participants) | 10
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0: number analyzed (Participants) | 10
  Protein: Day 121, 0 | 4
  Protein: Day 191, 0 | 4
  Protein: Day 191, 1+ | 2

8. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Day 15 and 29
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Participants
  Occult blood: 6 hours, 0 | 0
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 0
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 0
  Occult blood: 72 hours, 1+ | 0
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 0
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 0
  Occult blood: Day 29, 0 | 0
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 25 | 0
  Glucose: 6 hours, 0 | 0
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 0
  Glucose: 72 hours, 0 | 0
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 0
  Glucose: Day 15, 0 | 0
  Glucose: Day 29, 0 | 0
  Ketones: 6 hours, 0 | 0
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 0
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 0
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 0
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 0
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 29, 0 | 0
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 29, 1+ | 0
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 0
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 0
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 0
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 0
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 0
  Protein: Day 15, 1+ | 0
  Protein: Day 29, 0 | 0
  Protein: Day 29, 1+ | 0

9. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 29 and 43
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Participants
  Occult blood: 6 hours, 0 | 0
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 0
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 0
  Occult blood: 72 hours, 1+ | 0
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 0
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 0
  Occult blood: Day 29, 0 | 0
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 2+ | 0
  Occult blood: Day 29, 25 | 0
  Occult blood: Day 43, 0 | 0
  Occult blood: Day 43, 10 | 0
  Occult blood: Day 43, 25 | 0
  Glucose: 6 hours, 0 | 0
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 0
  Glucose: 72 hours, 0 | 0
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 0
  Glucose: Day 15, 0 | 0
  Glucose: Day 29, 0 | 0
  Glucose: Day 43, 0 | 0
  Ketones: 6 hours, 0 | 0
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 0
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 0
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 0
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 0
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 29, 0 | 0
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 43, 0 | 0
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1+ | 0
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 0
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 0
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 0
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 0
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 0
  Protein: Day 15, 1+ | 0
  Protein: Day 29, 0 | 0
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 0
  Protein: Day 43, 1+ | 0

10. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57 and 85
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, 0 | 0
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 0
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 0
  Occult blood: 72 hours, 1+ | 0
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 0
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 0
  Occult blood: Day 22, 0 | 0
  Occult blood: Day 22, 10 | 0
  Occult blood: Day 22, 2+ | 0
  Occult blood: Day 29, 0 | 0
  Occult blood: Day 29, 1+ | 0
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 2+ | 0
  Occult blood: Day 29, 25 | 0
  Occult blood: Day 43, 0 | 0
  Occult blood: Day 43, 1+ | 0
  Occult blood: Day 43, 10 | 0
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 57, 0 | 0
  Occult blood: Day 57, 1+ | 0
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 85, 0 | 0
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 85, 25 | 0
  Glucose: 6 hours, 0 | 0
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 0
  Glucose: 72 hours, 0 | 0
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 0
  Glucose: Day 15, 0 | 0
  Glucose: Day 22, 0 | 0
  Glucose: Day 29, 0 | 0
  Glucose: Day 43, 0 | 0
  Glucose: Day 57, 0 | 0
  Glucose: Day 85, 0 | 0
  Ketones: 6 hours, 0 | 0
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 0
  Ketones: 12 hours, 1+ | 1
  Ketones: 72 hours, 0 | 0
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 0
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 0
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 22, 0 | 0
  Ketones: Day 22, 0.5 | 0
  Ketones: Day 29, 0 | 0
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 43, 0 | 0
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 0
  Ketones: Day 85, 0 | 0
  Ketones: Day 85, 0.5 | 0
  Ketones: Day 85, 1+ | 1
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 0
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 0
  Protein: 12 hours, 2+ | 1
  Protein: 72 hours, 0 | 0
  Protein: 72 hours, 1+ | 1
  Protein: 168 hours, 0 | 0
  Protein: 168 hours, 1+ | 1
  Protein: 168 hours, 2+ | 1
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 0
  Protein: Day 15, 1+ | 1
  Protein: Day 22, 0 | 0
  Protein: Day 22, 1+ | 1
  Protein: Day 29, 0 | 0
  Protein: Day 29, 1+ | 1
  Protein: Day 43, 0 | 0
  Protein: Day 43, 1+ | 0
  Protein: Day 57, 0 | 0
  Protein: Day 57, 1+ | 1
  Protein: Day 85, 0 | 0
  Protein: Day 85, 1+ | 0

11. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.04 mg/kg (ADA-ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 147
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, 0 | 1
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 1
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 1
  Occult blood: 72 hours, 1+ | 0
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 1
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 1
  Occult blood: Day 22, 0 | 1
  Occult blood: Day 22, 10 | 0
  Occult blood: Day 22, 2+ | 0
  Occult blood: Day 29, 0 | 1
  Occult blood: Day 29, 1+ | 0
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 2+ | 0
  Occult blood: Day 29, 25 | 0
  Occult blood: Day 43, 0 | 1
  Occult blood: Day 43, 1+ | 0
  Occult blood: Day 43, 10 | 0
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 57, 0 | 1
  Occult blood: Day 57, 1+ | 0
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 85, 0 | 1
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 121, 0 | 0
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10 | 1
  Occult blood: Day 147, 0 | 1
  Occult blood: Day 147, 10 | 0
  Occult blood: Day 147, 25 | 0
  Glucose: 6 hours, 0 | 1
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 1
  Glucose: 72 hours, 0 | 1
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 1
  Glucose: Day 15, 0 | 1
  Glucose: Day 22, 0 | 1
  Glucose: Day 29, 0 | 1
  Glucose: Day 43, 0 | 1
  Glucose: Day 57, 0 | 1
  Glucose: Day 85, 0 | 1
  Glucose: Day 121, 0 | 1
  Glucose: Day 147, 0 | 1
  Ketones: 6 hours, 0 | 1
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 1
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 1
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 1
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 1
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 22, 0 | 1
  Ketones: Day 22, 0.5 | 0
  Ketones: Day 29, 0 | 1
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 43, 0 | 1
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 1
  Ketones: Day 85, 0 | 1
  Ketones: Day 85, 0.5 | 0
  Ketones: Day 121, 0 | 1
  Ketones: Day 121, 0.5 | 0
  Ketones: Day 121, 2+ | 0
  Ketones: Day 147, 0 | 1
  Ketones: Day 147, 0.5 | 0
  Ketones: Day 147, 1+ | 0
  Nitrite: Day 15, positive | 0
  Nitrite: Day 85, positive | 0
  Nitrite: Day 121, positive | 0
  Protein: 6 hours, 0 | 1
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 1
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 1
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 1
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 1
  Protein: Day 15, 1+ | 0
  Protein: Day 22, 0 | 1
  Protein: Day 22, 1+ | 0
  Protein: Day 29, 0 | 1
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 1
  Protein: Day 43, 1+ | 0
  Protein: Day 57, 0 | 1
  Protein: Day 57, 1+ | 0
  Protein: Day 85, 0 | 1
  Protein: Day 85, 1+ | 1
  Protein: Day 121, 0 | 1
  Protein: Day 147, 0 | 1
  Protein: Day 147, 1+ | 0

12. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.15 mg/kg (ADA-ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 219
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, 0 | 4
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 3
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 1
  Occult blood: 72 hours, 0 | 1
  Occult blood: 72 hours, 1+ | 1
  Occult blood: 72 hours, 10 | 2
  Occult blood: 72 hours, 50 | 1
  Occult blood: 168 hours, 0 | 2
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 1
  Occult blood: 168 hours, 25 | 1
  Occult blood: Day 15, 0 | 4
  Occult blood: Day 22, 0 | 3
  Occult blood: Day 22, 10 | 1
  Occult blood: Day 22, 2+ | 0
  Occult blood: Day 29, 0 | 2
  Occult blood: Day 29, 1+ | 0
  Occult blood: Day 29, 10 | 1
  Occult blood: Day 29, 2+ | 0
  Occult blood: Day 29, 25 | 1
  Occult blood: Day 43, 0 | 2
  Occult blood: Day 43, 1+ | 1
  Occult blood: Day 43, 10 | 1
  Occult blood: Day 43, 25 | 1
  Occult blood: Day 57, 0 | 2
  Occult blood: Day 57, 1+ | 0
  Occult blood: Day 57, 10 | 2
  Occult blood: Day 85, 0 | 3
  Occult blood: Day 85, 10 | 1
  Occult blood: Day 121, 0 | 2
  Occult blood: Day 121, 1+ | 1
  Occult blood: Day 121, 10 | 2
  Occult blood: Day 219, 0 | 1
  Occult blood: Day 219, 10 | 2
  Occult blood: Day 219, 25 | 1
  Glucose: 6 hours, 0 | 4
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 4
  Glucose: 72 hours, 0 | 4
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 4
  Glucose: Day 15, 0 | 4
  Glucose: Day 22, 0 | 4
  Glucose: Day 29, 0 | 4
  Glucose: Day 43, 0 | 4
  Glucose: Day 57, 0 | 4
  Glucose: Day 85, 0 | 4
  Glucose: Day 121, 0 | 4
  Glucose: Day 219, 0 | 4
  Ketones: 6 hours, 0 | 4
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 4
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 2
  Ketones: 72 hours, 0.5 | 2
  Ketones: 168 hours, 0 | 3
  Ketones: 168 hours, 0.5 | 1
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 4
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 22, 0 | 3
  Ketones: Day 22, 0.5 | 1
  Ketones: Day 29, 0 | 3
  Ketones: Day 29, 0.5 | 1
  Ketones: Day 43, 0 | 3
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1.5 | 1
  Ketones: Day 57, 0 | 4
  Ketones: Day 85, 0 | 4
  Ketones: Day 85, 0.5 | 0
  Ketones: Day 121, 0 | 4
  Ketones: Day 121, 0.5 | 0
  Ketones: Day 121, 2+ | 0
  Ketones: Day 219, 0 | 3
  Ketones: Day 219, 0.5 | 1
  Ketones: Day 219, 1+ | 0
  Nitrite: Day 15, positive | 0
  Nitrite: Day 85, positive | 0
  Nitrite: Day 121, positive | 0
  Protein: 6 hours, 0 | 4
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 4
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 4
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 4
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 4
  Protein: Day 15, 1+ | 0
  Protein: Day 22, 0 | 4
  Protein: Day 22, 1+ | 0
  Protein: Day 29, 0 | 4
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 4
  Protein: Day 43, 1+ | 0
  Protein: Day 57, 0 | 4
  Protein: Day 57, 1+ | 0
  Protein: Day 85, 0 | 4
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0 | 4
  Protein: Day 219, 0 | 4
  Protein: Day 219, 1+ | 0

13. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.15 mg/kg (ADA+ve)
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 191
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, 0 | 4
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 7 | 0
  Occult blood: 12 hours, 0 | 4
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 72 hours, 0 | 4
  Occult blood: 72 hours, 1+ | 0
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 50 | 0
  Occult blood: 168 hours, 0 | 3
  Occult blood: 168 hours, 1+ | 0
  Occult blood: 168 hours, 10 | 1
  Occult blood: 168 hours, 25 | 0
  Occult blood: Day 15, 0 | 4
  Occult blood: Day 22, 0 | 4
  Occult blood: Day 22, 10 | 0
  Occult blood: Day 22, 2+ | 0
  Occult blood: Day 29, 0 | 4
  Occult blood: Day 29, 1+ | 0
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 2+ | 0
  Occult blood: Day 29, 25 | 0
  Occult blood: Day 43, 0 | 4
  Occult blood: Day 43, 1+ | 0
  Occult blood: Day 43, 10 | 0
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 57, 0 | 4
  Occult blood: Day 57, 1+ | 0
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 85, 0 | 4
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 121, 0 | 4
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10 | 0
  Occult blood: Day 191, 0 | 4
  Occult blood: Day 191, 10 | 0
  Occult blood: Day 191, 25 | 0
  Glucose: 6 hours, 0 | 4
  Glucose: 6 hours, 17 | 0
  Glucose: 6 hours, 7 | 0
  Glucose: 12 hours, 0 | 4
  Glucose: 72 hours, 0 | 4
  Glucose: 72 hours, 3 | 0
  Glucose: 168 hours, 0 | 4
  Glucose: Day 15, 0 | 4
  Glucose: Day 22, 0 | 4
  Glucose: Day 29, 0 | 4
  Glucose: Day 43, 0 | 4
  Glucose: Day 57, 0 | 4
  Glucose: Day 85, 0 | 4
  Glucose: Day 121, 0 | 4
  Glucose: Day 191, 0 | 4
  Ketones: 6 hours, 0 | 4
  Ketones: 6 hours, 7 | 0
  Ketones: 12 hours, 0 | 4
  Ketones: 12 hours, 1+ | 0
  Ketones: 72 hours, 0 | 4
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 4
  Ketones: 168 hours, 0.5 | 0
  Ketones: 168 hours, 4+ | 0
  Ketones: Day 15, 0 | 4
  Ketones: Day 15, 0.5 | 0
  Ketones: Day 22, 0 | 4
  Ketones: Day 22, 0.5 | 0
  Ketones: Day 29, 0 | 2
  Ketones: Day 29, 0.5 | 2
  Ketones: Day 43, 0 | 3
  Ketones: Day 43, 0.5 | 1
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 4
  Ketones: Day 85, 0 | 3
  Ketones: Day 85, 0.5 | 1
  Ketones: Day 121, 0 | 3
  Ketones: Day 121, 0.5 | 1
  Ketones: Day 121, 2+ | 0
  Ketones: Day 191, 0 | 4
  Ketones: Day 191, 0.5 | 0
  Ketones: Day 191, 1+ | 0
  Nitrite: Day 15, positive | 0
  Nitrite: Day 85, positive | 0
  Nitrite: Day 121, positive | 0
  Protein: 6 hours, 0 | 4
  Protein: 6 hours, 7 | 0
  Protein: 12 hours, 0 | 4
  Protein: 12 hours, 2+ | 0
  Protein: 72 hours, 0 | 4
  Protein: 72 hours, 1+ | 0
  Protein: 168 hours, 0 | 4
  Protein: 168 hours, 1+ | 0
  Protein: 168 hours, 2+ | 0
  Protein: 168 hours, 3+ | 0
  Protein: Day 15, 0 | 4
  Protein: Day 15, 1+ | 0
  Protein: Day 22, 0 | 4
  Protein: Day 22, 1+ | 0
  Protein: Day 29, 0 | 4
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 4
  Protein: Day 43, 1+ | 0
  Protein: Day 57, 0 | 4
  Protein: Day 57, 1+ | 0
  Protein: Day 85, 0 | 4
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0 | 4
  Protein: Day 191, 0 | 4
  Protein: Day 191, 1+ | 0

14. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for Psoriasis Placebo
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 307
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Psoriasis
Number analyzed (Participants) | 9
Participants
  Occult blood: 6 hours, + | 1
  Occult blood: 6 hours, 0 | 4
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 2
  Occult blood: 6 hours, 50 | 0
  Occult blood: 12 hours, + | 1
  Occult blood: 12 hours, 0 | 3
  Occult blood: 12 hours, 10 | 0
  Occult blood: 12 hours, 150 | 0
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 2
  Occult blood: 12 hours, 50 | 1
  Occult blood: 72 hours, + | 1
  Occult blood: 72 hours, 0 | 2
  Occult blood: 72 hours, 10 | 2
  Occult blood: 72 hours, 150 | 1
  Occult blood: 72 hours, 25 | 1
  Occult blood: 168 hours, 0 | 4
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 150 | 1
  Occult blood: 168 hours, 25 | 1
  Occult blood: 168 hours, 250 | 0
  Occult blood: Day 15, 0 | 3
  Occult blood: Day 15, 10 | 1
  Occult blood: Day 15, 25 | 1
  Occult blood: Day 15, 250 | 0
  Occult blood: Day 15, 50 | 1
  Occult blood: Day 22, 0 | 3
  Occult blood: Day 22, 1+ | 0
  Occult blood: Day 22, 10 | 1
  Occult blood: Day 22, 150 | 0
  Occult blood: Day 22, 25 | 1
  Occult blood: Day 22, 50 | 1
  Occult blood: Day 29, 0 | 4
  Occult blood: Day 29, 10 | 1
  Occult blood: Day 29, 150 | 0
  Occult blood: Day 29, 50 | 1
  Occult blood: Day 43, 0 | 2
  Occult blood: Day 43, 10 | 2
  Occult blood: Day 43, 150 | 0
  Occult blood: Day 43, 25 | 1
  Occult blood: Day 43, 3+ | 0
  Occult blood: Day 43, 50 | 1
  Occult blood: Day 57, 0 | 3
  Occult blood: Day 57, 10 | 1
  Occult blood: Day 57, 150 | 0
  Occult blood: Day 57, 25 | 1
  Occult blood: Day 57, 50 | 1
  Occult blood: Day 85, 0 | 4
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 85, 25 | 1
  Occult blood: Day 85, 50 | 1
  Occult blood: Day 121, + | 1
  Occult blood: Day 121, 0 | 4
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10 | 0
  Occult blood: Day 121, 150 | 0
  Occult blood: Day 121, 25 | 2
  Occult blood: Day 307, 0 | 3
  Occult blood: Day 307, 10 | 0
  Occult blood: Day 307, 25 | 2
  Occult blood: Day 307, 50 | 1
  Glucose: 6 hours, 0 | 6
  Glucose: 12 hours, 0 | 5
  Glucose: 12 hours, 9 | 1
  Glucose: 72 hours, 0 | 6
  Glucose: 168 hours, 0 | 6
  Glucose: Day 15, 0 | 6
  Glucose: Day 22, 0 | 6
  Glucose: Day 22, 5 | 0
  Glucose: Day 29, 0 | 6
  Glucose: Day 43, 0 | 6
  Glucose: Day 57, 0 | 6
  Glucose: Day 85, 0 | 6
  Glucose: Day 121, 0 | 6
  Glucose: Day 307, 0 | 6
  Ketones: 6 hours, 0 | 6
  Ketones: 12 hours, 0 | 5
  Ketones: 12 hours, 0.5 | 1
  Ketones: 72 hours, 0 | 6
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 5
  Ketones: 168 hours, 0.5 | 1
  Ketones: Day 15, 0 | 4
  Ketones: Day 15, 0.5 | 2
  Ketones: Day 22, 0 | 5
  Ketones: Day 22, 0.5 | 1
  Ketones: Day 29, 0 | 5
  Ketones: Day 29, 0.5 | 1
  Ketones: Day 43, 0 | 5
  Ketones: Day 43, 0.5 | 1
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 5
  Ketones: Day 57, 0.5 | 1
  Ketones: Day 85, 0 | 5
  Ketones: Day 85, 0.5 | 1
  Ketones: Day 121, 0 | 4
  Ketones: Day 121, 0.5 | 2
  Ketones: Day 307, 0 | 5
  Ketones: Day 307, 0.5 | 1
  Nitrite: Day 15, positive | 1
  Protein: 6 hours, 0 | 6
  Protein: 12 hours, 0 | 6
  Protein: 72 hours, 0 | 6
  Protein: 168 hours, 0 | 6
  Protein: 168 hours, 0.25 | 0
  Protein: 168 hours, 1+ | 1
  Protein: Day 15, 0 | 6
  Protein: Day 15, 0.25 | 0
  Protein: Day 22, 0 | 6
  Protein: Day 22, 0.25 | 0
  Protein: Day 29, 0 | 5
  Protein: Day 29, 0.25 | 1
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 6
  Protein: Day 43, 0.25 | 0
  Protein: Day 57, 0 | 6
  Protein: Day 85, 0 | 6
  Protein: Day 85, 0.25 | 0
  Protein: Day 85, 1+ | 1
  Protein: Day 121, 0 | 6
  Protein: Day 307, 0 | 6
  Protein: Day 307, 0.25 | 0

15. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 0.5 mg/kg
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 237
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, + | 0
  Occult blood: 6 hours, 0 | 2
  Occult blood: 6 hours, 1+ | 1
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 50 | 0
  Occult blood: 12 hours, + | 0
  Occult blood: 12 hours, 0 | 2
  Occult blood: 12 hours, 10 | 0
  Occult blood: 12 hours, 150 | 0
  Occult blood: 12 hours, 2+ | 1
  Occult blood: 12 hours, 25 | 0
  Occult blood: 12 hours, 50 | 0
  Occult blood: 72 hours, + | 0
  Occult blood: 72 hours, 0 | 2
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 150 | 0
  Occult blood: 72 hours, 25 | 0
  Occult blood: 168 hours, 0 | 2
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 150 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: 168 hours, 250 | 0
  Occult blood: Day 15, 0 | 2
  Occult blood: Day 15, 10 | 0
  Occult blood: Day 15, 25 | 0
  Occult blood: Day 15, 250 | 0
  Occult blood: Day 15, 50 | 0
  Occult blood: Day 22, 0 | 2
  Occult blood: Day 22, 1+ | 1
  Occult blood: Day 22, 10 | 0
  Occult blood: Day 22, 150 | 0
  Occult blood: Day 22, 25 | 0
  Occult blood: Day 22, 50 | 0
  Occult blood: Day 29, 0 | 2
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 150 | 0
  Occult blood: Day 29, 50 | 0
  Occult blood: Day 43, 0 | 1
  Occult blood: Day 43, 10 | 1
  Occult blood: Day 43, 150 | 0
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 43, 3+ | 1
  Occult blood: Day 43, 50 | 0
  Occult blood: Day 57, 0 | 2
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 57, 150 | 0
  Occult blood: Day 57, 25 | 0
  Occult blood: Day 57, 50 | 0
  Occult blood: Day 85, 0 | 2
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 85, 25 | 0
  Occult blood: Day 85, 50 | 0
  Occult blood: Day 121, + | 0
  Occult blood: Day 121, 0 | 2
  Occult blood: Day 121, 1+ | 1
  Occult blood: Day 121, 10 | 0
  Occult blood: Day 121, 150 | 0
  Occult blood: Day 121, 25 | 0
  Occult blood: Day 237, 0 | 2
  Occult blood: Day 237, 10 | 0
  Occult blood: Day 237, 25 | 0
  Occult blood: Day 237, 50 | 0
  Glucose: 6 hours, 0 | 2
  Glucose: 12 hours, 0 | 2
  Glucose: 12 hours, 9 | 0
  Glucose: 72 hours, 0 | 2
  Glucose: 168 hours, 0 | 2
  Glucose: Day 15, 0 | 2
  Glucose: Day 22, 0 | 2
  Glucose: Day 22, 5 | 0
  Glucose: Day 29, 0 | 2
  Glucose: Day 43, 0 | 2
  Glucose: Day 57, 0 | 2
  Glucose: Day 85, 0 | 2
  Glucose: Day 121, 0 | 2
  Glucose: Day 237, 0 | 2
  Ketones: 6 hours, 0 | 2
  Ketones: 12 hours, 0 | 2
  Ketones: 12 hours, 0.5 | 0
  Ketones: 72 hours, 0 | 2
  Ketones: 72 hours, 0.5 | 0
  Ketones: 168 hours, 0 | 2
  Ketones: 168 hours, 0.5 | 0
  Ketones: Day 15, 0 | 0
  Ketones: Day 15, 0.5 | 2
  Ketones: Day 22, 0 | 1
  Ketones: Day 22, 0.5 | 1
  Ketones: Day 29, 0 | 1
  Ketones: Day 29, 0.5 | 1
  Ketones: Day 43, 0 | 1
  Ketones: Day 43, 0.5 | 1
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 6
  Ketones: Day 57, 0.5 | 0
  Ketones: Day 85, 0 | 2
  Ketones: Day 85, 0.5 | 0
  Ketones: Day 121, 0 | 1
  Ketones: Day 121, 0.5 | 1
  Ketones: Day 237, 0 | 2
  Ketones: Day 237, 0.5 | 0
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 2
  Protein: 12 hours, 0 | 2
  Protein: 72 hours, 0 | 2
  Protein: 168 hours, 0 | 2
  Protein: 168 hours, 0.25 | 0
  Protein: 168 hours, 1+ | 0
  Protein: Day 15, 0 | 2
  Protein: Day 15, 0.25 | 0
  Protein: Day 22, 0 | 2
  Protein: Day 22, 0.25 | 0
  Protein: Day 29, 0 | 2
  Protein: Day 29, 0.25 | 0
  Protein: Day 29, 1+ | 1
  Protein: Day 43, 0 | 2
  Protein: Day 43, 0.25 | 0
  Protein: Day 57, 0 | 2
  Protein: Day 85, 0 | 2
  Protein: Day 85, 0.25 | 0
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0 | 2
  Protein: Day 237, 0 | 2
  Protein: Day 237, 0.25 | 0

16. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 1.5 mg/kg
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 277
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, + | 0
  Occult blood: 6 hours, 0 | 4
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 1
  Occult blood: 6 hours, 50 | 1
  Occult blood: 12 hours, + | 0
  Occult blood: 12 hours, 0 | 5
  Occult blood: 12 hours, 10 | 0
  Occult blood: 12 hours, 150 | 1
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 12 hours, 50 | 0
  Occult blood: 72 hours, + | 0
  Occult blood: 72 hours, 0 | 4
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 150 | 1
  Occult blood: 72 hours, 25 | 1
  Occult blood: 168 hours, 0 | 4
  Occult blood: 168 hours, 10 | 1
  Occult blood: 168 hours, 150 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: 168 hours, 250 | 1
  Occult blood: Day 15, 0 | 4
  Occult blood: Day 15, 10 | 1
  Occult blood: Day 15, 25 | 0
  Occult blood: Day 15, 250 | 1
  Occult blood: Day 15, 50 | 0
  Occult blood: Day 22, 0 | 4
  Occult blood: Day 22, 1+ | 0
  Occult blood: Day 22, 10 | 1
  Occult blood: Day 22, 150 | 1
  Occult blood: Day 22, 25 | 0
  Occult blood: Day 22, 50 | 0
  Occult blood: Day 29, 0 | 3
  Occult blood: Day 29, 10 | 2
  Occult blood: Day 29, 150 | 1
  Occult blood: Day 29, 50 | 0
  Occult blood: Day 43, 0 | 3
  Occult blood: Day 43, 10 | 1
  Occult blood: Day 43, 150 | 1
  Occult blood: Day 43, 25 | 1
  Occult blood: Day 43, 3+ | 0
  Occult blood: Day 43, 50 | 0
  Occult blood: Day 57, 0 | 4
  Occult blood: Day 57, 10 | 1
  Occult blood: Day 57, 150 | 1
  Occult blood: Day 57, 25 | 0
  Occult blood: Day 57, 50 | 0
  Occult blood: Day 85, 0 | 5
  Occult blood: Day 85, 10 | 0
  Occult blood: Day 85, 25 | 1
  Occult blood: Day 85, 50 | 0
  Occult blood: Day 121, + | 0
  Occult blood: Day 121, 0 | 4
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10 | 1
  Occult blood: Day 121, 150 | 1
  Occult blood: Day 121, 25 | 0
  Occult blood: Day 277, 0 | 4
  Occult blood: Day 277, 10 | 0
  Occult blood: Day 277, 25 | 1
  Occult blood: Day 277, 50 | 1
  Glucose: 6 hours, 0 | 6
  Glucose: 12 hours, 0 | 6
  Glucose: 12 hours, 9 | 0
  Glucose: 72 hours, 0 | 6
  Glucose: 168 hours, 0 | 6
  Glucose: Day 15, 0 | 6
  Glucose: Day 22, 0 | 5
  Glucose: Day 22, 5 | 1
  Glucose: Day 29, 0 | 6
  Glucose: Day 43, 0 | 6
  Glucose: Day 57, 0 | 6
  Glucose: Day 85, 0 | 6
  Glucose: Day 121, 0 | 6
  Glucose: Day 277, 0 | 6
  Ketones: 6 hours, 0 | 6
  Ketones: 12 hours, 0 | 6
  Ketones: 12 hours, 0.5 | 0
  Ketones: 72 hours, 0 | 5
  Ketones: 72 hours, 0.5 | 1
  Ketones: 168 hours, 0 | 6
  Ketones: 168 hours, 0.5 | 0
  Ketones: Day 15, 0 | 5
  Ketones: Day 15, 0.5 | 1
  Ketones: Day 22, 0 | 4
  Ketones: Day 22, 0.5 | 2
  Ketones: Day 29, 0 | 5
  Ketones: Day 29, 0.5 | 1
  Ketones: Day 43, 0 | 5
  Ketones: Day 43, 0.5 | 0
  Ketones: Day 43, 1.5 | 1
  Ketones: Day 57, 0 | 5
  Ketones: Day 57, 0.5 | 1
  Ketones: Day 85, 0 | 6
  Ketones: Day 85, 0.5 | 0
  Ketones: Day 121, 0 | 6
  Ketones: Day 121, 0.5 | 0
  Ketones: Day 277, 0 | 6
  Ketones: Day 277, 0.5 | 0
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 6
  Protein: 12 hours, 0 | 6
  Protein: 72 hours, 0 | 6
  Protein: 168 hours, 0 | 5
  Protein: 168 hours, 0.25 | 1
  Protein: 168 hours, 1+ | 0
  Protein: Day 15, 0 | 5
  Protein: Day 15, 0.25 | 1
  Protein: Day 22, 0 | 4
  Protein: Day 22, 0.25 | 2
  Protein: Day 29, 0 | 6
  Protein: Day 29, 0.25 | 0
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 5
  Protein: Day 43, 0.25 | 1
  Protein: Day 57, 0 | 6
  Protein: Day 85, 0 | 5
  Protein: Day 85, 0.25 | 1
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0 | 6
  Protein: Day 277, 0 | 5
  Protein: Day 277, 0.25 | 1

17. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick for GSK2831781 5 mg/kg
Description: as for outcome 7
Time Frame: 6, 12, 72, 168 hours, Days 15, 22, 29, 43, 57, 85, 121 and 307
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
Participants
  Occult blood: 6 hours, + | 0
  Occult blood: 6 hours, 0 | 5
  Occult blood: 6 hours, 1+ | 0
  Occult blood: 6 hours, 10 | 0
  Occult blood: 6 hours, 50 | 0
  Occult blood: 12 hours, + | 0
  Occult blood: 12 hours, 0 | 4
  Occult blood: 12 hours, 10 | 1
  Occult blood: 12 hours, 150 | 0
  Occult blood: 12 hours, 2+ | 0
  Occult blood: 12 hours, 25 | 0
  Occult blood: 12 hours, 50 | 0
  Occult blood: 72 hours, + | 0
  Occult blood: 72 hours, 0 | 5
  Occult blood: 72 hours, 10 | 0
  Occult blood: 72 hours, 150 | 0
  Occult blood: 72 hours, 25 | 0
  Occult blood: 168 hours, 0 | 5
  Occult blood: 168 hours, 10 | 0
  Occult blood: 168 hours, 150 | 0
  Occult blood: 168 hours, 25 | 0
  Occult blood: 168 hours, 250 | 0
  Occult blood: Day 15, 0 | 5
  Occult blood: Day 15, 10 | 0
  Occult blood: Day 15, 25 | 0
  Occult blood: Day 15, 250 | 0
  Occult blood: Day 15, 50 | 0
  Occult blood: Day 22, 0: number analyzed (Participants) | 5
  Occult blood: Day 22, 0 | 4
  Occult blood: Day 22, 1+: number analyzed (Participants) | 5
  Occult blood: Day 22, 1+ | 0
  Occult blood: Day 22, 10: number analyzed (Participants) | 5
  Occult blood: Day 22, 10 | 1
  Occult blood: Day 22, 150: number analyzed (Participants) | 5
  Occult blood: Day 22, 150 | 0
  Occult blood: Day 22, 25: number analyzed (Participants) | 5
  Occult blood: Day 22, 25 | 0
  Occult blood: Day 22, 50: number analyzed (Participants) | 5
  Occult blood: Day 22, 50 | 0
  Occult blood: Day 29, 0 | 5
  Occult blood: Day 29, 10 | 0
  Occult blood: Day 29, 150 | 0
  Occult blood: Day 29, 50 | 0
  Occult blood: Day 43, 0 | 4
  Occult blood: Day 43, 10 | 1
  Occult blood: Day 43, 150 | 0
  Occult blood: Day 43, 25 | 0
  Occult blood: Day 43, 3+ | 0
  Occult blood: Day 43, 50 | 0
  Occult blood: Day 57, 0 | 5
  Occult blood: Day 57, 10 | 0
  Occult blood: Day 57, 150 | 0
  Occult blood: Day 57, 25 | 0
  Occult blood: Day 57, 50 | 0
  Occult blood: Day 85, 0 | 4
  Occult blood: Day 85, 10 | 1
  Occult blood: Day 85, 25 | 0
  Occult blood: Day 85, 50 | 0
  Occult blood: Day 121, + | 0
  Occult blood: Day 121, 0 | 4
  Occult blood: Day 121, 1+ | 0
  Occult blood: Day 121, 10 | 1
  Occult blood: Day 121, 150 | 0
  Occult blood: Day 121, 25 | 0
  Occult blood: Day 307, 0 | 4
  Occult blood: Day 307, 10 | 1
  Occult blood: Day 307, 25 | 0
  Occult blood: Day 307, 50 | 0
  Glucose: 6 hours, 0 | 5
  Glucose: 12 hours, 0 | 5
  Glucose: 12 hours, 9 | 0
  Glucose: 72 hours, 0 | 5
  Glucose: 168 hours, 0 | 5
  Glucose: Day 15, 0 | 5
  Glucose: Day 22, 0: number analyzed (Participants) | 5
  Glucose: Day 22, 0 | 5
  Glucose: Day 22, 5: number analyzed (Participants) | 5
  Glucose: Day 22, 5 | 0
  Glucose: Day 29, 0 | 5
  Glucose: Day 43, 0 | 5
  Glucose: Day 57, 0 | 5
  Glucose: Day 85, 0 | 5
  Glucose: Day 121, 0 | 5
  Glucose: Day 307, 0 | 5
  Ketones: 6 hours, 0 | 5
  Ketones: 12 hours, 0 | 4
  Ketones: 12 hours, 0.5 | 1
  Ketones: 72 hours, 0 | 4
  Ketones: 72 hours, 0.5 | 1
  Ketones: 168 hours, 0 | 3
  Ketones: 168 hours, 0.5 | 2
  Ketones: Day 15, 0 | 4
  Ketones: Day 15, 0.5 | 1
  Ketones: Day 22, 0: number analyzed (Participants) | 5
  Ketones: Day 22, 0 | 5
  Ketones: Day 22, 0.5: number analyzed (Participants) | 5
  Ketones: Day 22, 0.5 | 0
  Ketones: Day 29, 0 | 5
  Ketones: Day 29, 0.5 | 0
  Ketones: Day 43, 0 | 3
  Ketones: Day 43, 0.5 | 2
  Ketones: Day 43, 1.5 | 0
  Ketones: Day 57, 0 | 4
  Ketones: Day 57, 0.5 | 1
  Ketones: Day 85, 0 | 3
  Ketones: Day 85, 0.5 | 2
  Ketones: Day 121, 0 | 3
  Ketones: Day 121, 0.5 | 2
  Ketones: Day 307, 0 | 5
  Ketones: Day 307, 0.5 | 0
  Nitrite: Day 15, positive | 0
  Protein: 6 hours, 0 | 5
  Protein: 12 hours, 0 | 5
  Protein: 72 hours, 0 | 5
  Protein: 168 hours, 0 | 5
  Protein: 168 hours, 0.25 | 0
  Protein: 168 hours, 1+ | 0
  Protein: Day 15, 0 | 5
  Protein: Day 15, 0.25 | 0
  Protein: Day 22, 0: number analyzed (Participants) | 5
  Protein: Day 22, 0 | 5
  Protein: Day 22, 0.25: number analyzed (Participants) | 5
  Protein: Day 22, 0.25 | 0
  Protein: Day 29, 0 | 5
  Protein: Day 29, 0.25 | 0
  Protein: Day 29, 1+ | 0
  Protein: Day 43, 0 | 5
  Protein: Day 43, 0.25 | 0
  Protein: Day 57, 0 | 5
  Protein: Day 85, 0 | 5
  Protein: Day 85, 0.25 | 0
  Protein: Day 85, 1+ | 0
  Protein: Day 121, 0 | 5
  Protein: Day 307, 0 | 5
  Protein: Day 307, 0.25 | 0

18. Secondary Outcome: Change From Baseline (PPD First Challenge) of Induration Diameter From Re-challenge at 3 Days Post-dose
Description: The induration diameter by challenge site is defined as the average of the two skin response test values (vertical and horizontal) at each challenge site. A challenge site is defined by skin response (SR) directionality (upper/lower) and SR laterality (left/right). Four categories considered were as follows: left upper, right upper, left lower and right lower. Baseline was considered as Day -26. Change from Baseline was calculated as post-Baseline value minus Baseline value. Data is presented for DTH participants.
Time Frame: Baseline, Days 4, 8, 15 and 22 post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Groups:
- Placebo for Healthy Volunteer: Healthy volunteers with DTH received a single dose of placebo-matching saline solution, intravenously on Day 1 for 2 hours post-infusion start.
Arm/Group | Placebo for Healthy Volunteer | GSK2831781 0.15 mg/kg (ADA-ve)
Number analyzed (Participants) | 6 | 6
Millimeter (mm)
  Day 4: Left upper average (n=6,6) | 3.167 (1.8886) | 6.500 (4.5497)
  Day 4: Right upper average (n=6,6) | 2.000 (4.2426) | 6.500 (4.3359)
  Day 8: Left upper average (n=5,3): number analyzed (Participants) | 5 | 3
  Day 8: Left upper average (n=5,3) | 0.300 (4.4805) | 2.167 (5.0083)
  Day 8: Right upper average (n=6,5): number analyzed (Participants) | 6 | 5
  Day 8: Right upper average (n=6,5) | -0.917 (7.8065) | -0.700 (4.2367)
  Day 15: Left upper average (n=5,3): number analyzed (Participants) | 5 | 3
  Day 15: Left upper average (n=5,3) | -7.500 (10.9430) | -3.333 (7.2342)
  Day 15: Right upper average (n=6,5): number analyzed (Participants) | 6 | 5
  Day 15: Right upper average (n=6,5) | -9.000 (9.8894) | -5.800 (2.9283)
  Day 22: Left upper average (n=5,3): number analyzed (Participants) | 5 | 3
  Day 22: Left upper average (n=5,3) | -11.600 (8.9121) | -11.833 (7.1122)
  Day 22: Right upper average (n=6,5): number analyzed (Participants) | 6 | 5
  Day 22: Right upper average (n=6,5) | -14.083 (10.4231) | -8.900 (9.7877)

19. Secondary Outcome: Duration of Induration in the Re-challenge for DTH
Description: The duration of induration was the time (in days) to achieve an overall induration less than 6 mm from the time of the PPD re-challenge post-dose. Duration of induration was calculated as: PPD re-challenge post-dose up to the last available induration measurement. Data is presented for DTH participants.
Time Frame: Up to 28 days post-dose
Population: Safety population.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo for Healthy Volunteer | GSK2831781 0.15 mg/kg (ADA-ve)
Number analyzed (Participants) | 6 | 6
Days | 20.0 [13 to 22] | 20.0 [13 to 21]

20. Secondary Outcome: Change From Baseline (PPD First Challenge) of Lymphocyte Activation Gene-3 (LAG-3)+ Cells in Biopsies of Re-challenged Skin at 3 Days Post-dose
Description: A punch biopsy was taken from one of the challenge sites. Cells in biopsies of re-challenged skin were measured by immunohistochemistry (IHC) and the LAG-3+ cells characterized and counted. Baseline was considered as Day -26 for this outcome measure. Change from Baseline was calculated as post-Baseline value minus Baseline value. Data is presented for DTH participants.
Time Frame: Baseline and 72 hours post-dose
Population: Safety population.
Measure: Mean (Standard Deviation); unit: LAG3+ cells
Arm/Group | Placebo for Healthy Volunteer | GSK2831781 0.15 mg/kg (ADA-ve)
Number analyzed (Participants) | 6 | 6
LAG3+ cells | 15.3 (24.90) | 19.7 (18.10)

21. Secondary Outcome: Change From Baseline in LAG-3+ Cells in Lesional Biopsies in Psoriasis Participants at Day 29
Description: A punch biopsy was taken from active leading edge of the lesion. Cells in lesional biopsies of skin were measured by IHC and count the LAG-3+ cells. The regions of interest for LAG3+ were located in epidermis and dermis. Baseline was considered as the latest pre-dose assessment with a non-missing value for Day -1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline and Day 29
Population: Safety population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: LAG3+ cells
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
LAG3+ cells
  Skin: Dermis (n=6,4,3,4): number analyzed (Participants) | 6 | 4 | 3 | 4
  Skin: Dermis (n=6,4,3,4) | 2.7 (6.09) | -2.5 (3.70) | 0.3 (2.08) | -2.5 (2.38)
  Skin: Epidermis (n=6,4,4,5): number analyzed (Participants) | 6 | 4 | 4 | 5
  Skin: Epidermis (n=6,4,4,5) | -1.2 (12.86) | -9.8 (15.11) | -6.5 (6.45) | -5.0 (6.89)

22. Secondary Outcome: Area Under the Plasma Time Curve From Zero to Infinity (AUC[0-infinity]) of GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma. Pharmacokinetic (PK) population consisted of all participants in the Safety Population who had at least 1 non-missing PK assessment.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for AUC(0-infinity) as there were not enough data points collected for a terminal slope required to calculate AUC(0-infinity).
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

23. Secondary Outcome: AUC(0-infinity) for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

24. Secondary Outcome: AUC(0-infinity) for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

25. Secondary Outcome: AUC(0-infinity) for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

26. Secondary Outcome: AUC(0-infinity) for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: AUC(0-infinity) for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

28. Secondary Outcome: AUC(0-infinity) for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

29. Secondary Outcome: AUC(0-infinity) for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 22
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

30. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-t]) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data was not collected because none of the participants had data evaluable for this measure.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

31. Secondary Outcome: AUC(0-t) for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
h*mcg/mL | 0.0060 (NA) — Geometric coefficient of variation could not be calculated for one participant.

32. Secondary Outcome: AUC(0-t) for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
h*mcg/mL | 1.3497 (31.95218)

33. Secondary Outcome: AUC(0-t) for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
h*mcg/mL | 23.6008 (27.26266)

34. Secondary Outcome: AUC(0-t) for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6 | 6
h*mcg/mL | 168.3458 (18.00654) | 238.1434 (43.68332)

35. Secondary Outcome: AUC(0-t) for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | 1187.8496 (34.15549)

36. Secondary Outcome: AUC(0-t) for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | 8493.7344 (13.62279)

37. Secondary Outcome: AUC(0-t) for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | 40599.8938 (23.74167)

38. Secondary Outcome: Area Under the Concentration-time Curve From Zero (Pre-dose) to Week 4 (AUC[0-Week 4]) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24 and 696 (Week 4) hours post-dose
Population: PK population. Data was not collected because none of the participants had data evaluable for this measure.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

39. Secondary Outcome: AUC(0-Week 4) for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 696 (Week 4) hours post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

40. Secondary Outcome: AUC(0-Week 4) for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

41. Secondary Outcome: AUC(0-Week 4) for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time point for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

42. Secondary Outcome: AUC(0-Week 4) for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6 | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC. | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

43. Secondary Outcome: AUC(0-Week 4) for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

44. Secondary Outcome: AUC(0-Week 4) for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time point for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

45. Secondary Outcome: AUC(0-Week 4) for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22 and 29 (Week 4) post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
h*mcg/mL | NA (NA) — As per predefined analysis plan,AUC(0-Week4) was not derived:concentrations dropped below limit of quantification before Week4, extrapolation was not possible as half-life could not be derived.Instead,AUC(0-t) describe total exposure in terms of AUC.

46. Secondary Outcome: Percentage of AUC(0-infinity) Obtained by Extrapolation (%AUCex) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for %AUCex as there were not enough data points collected for a terminal slope required to calculate %AUCex.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

47. Secondary Outcome: %AUCex for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

48. Secondary Outcome: %AUCex for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

49. Secondary Outcome: %AUCex for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

50. Secondary Outcome: %AUCex for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: %AUCex for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

52. Secondary Outcome: %AUCex for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

53. Secondary Outcome: %AUCex for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 46
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

54. Secondary Outcome: Maximum Observed Concentration (Cmax) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
mcg/mL | NA (NA) — Data could not be analyzed because data was below the limit of quantitation.

55. Secondary Outcome: Cmax for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
mcg/mL | 0.0127 (NA) — Geometric coefficient of variation could not be calculated for one participant.

56. Secondary Outcome: Cmax for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
mcg/mL | 0.1523 (19.07315)

57. Secondary Outcome: Cmax for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
mcg/mL | 0.8196 (25.57947)

58. Secondary Outcome: Cmax for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6 | 6
mcg/mL | 3.0047 (17.41022) | 3.4255 (18.07808)

59. Secondary Outcome: Cmax for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
mcg/mL | 8.4810 (23.51712)

60. Secondary Outcome: Cmax for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
mcg/mL | 41.1481 (15.53659)

61. Secondary Outcome: Cmax for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
mcg/mL | 158.8243 (22.22170)

62. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Hours | NA [NA to NA] — Data could not be analyzed because data was below the limit of quantitation.

63. Secondary Outcome: Tmax for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Hours | 1.950 [1.95 to 1.95]

64. Secondary Outcome: Tmax for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Hours | 1.950 [1.87 to 3.98]

65. Secondary Outcome: Tmax for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Hours | 4.025 [1.90 to 11.98]

66. Secondary Outcome: Tmax for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6 | 6
Hours | 1.980 [1.87 to 8.00] | 4.990 [1.95 to 8.07]

67. Secondary Outcome: Tmax for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
Hours | 3.930 [1.95 to 8.02]

68. Secondary Outcome: Tmax for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
Hours | 1.990 [1.93 to 4.40]

69. Secondary Outcome: Tmax for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
Hours | 2.975 [1.95 to 71.82]

70. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data was not collected because none of the participants had data evaluable for this measure.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

71. Secondary Outcome: Tlast for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Hours | 1.950 [1.95 to 1.95]

72. Secondary Outcome: Tlast for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Hours | 18.005 [12.02 to 24.30]

73. Secondary Outcome: Tlast for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Hours | 72.065 [47.92 to 72.38]

74. Secondary Outcome: Tlast for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6 | 6
Hours | 238.750 [165.00 to 241.02] | 288.235 [144.10 to 407.68]

75. Secondary Outcome: Tlast for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
Hours | 468.655 [314.00 to 507.07]

76. Secondary Outcome: Tlast for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
Hours | 1343.930 [1003.55 to 1345.02]

77. Secondary Outcome: Tlast for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
Hours | 2016.050 [1677.67 to 2042.30]

78. Secondary Outcome: Systemic Clearance of Parent Drug (CL) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for CL as there were not enough data points collected for a terminal slope required to calculate CL.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

79. Secondary Outcome: CL for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

80. Secondary Outcome: CL for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

81. Secondary Outcome: CL for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

82. Secondary Outcome: CL for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

83. Secondary Outcome: CL for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

84. Secondary Outcome: CL for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

85. Secondary Outcome: CL for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 78
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

86. Secondary Outcome: Volume of Distribution at Steady State (Vss) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for Vss as there were not enough data points collected for a terminal slope required to calculate Vss.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

87. Secondary Outcome: Vss for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

88. Secondary Outcome: Vss for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

89. Secondary Outcome: Vss for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

90. Secondary Outcome: Vss for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

91. Secondary Outcome: Vss for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

92. Secondary Outcome: Vss for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

93. Secondary Outcome: Vss for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 86
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

94. Secondary Outcome: Mean Residence Time (MRT) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for MRT as there were not enough data points collected for a terminal slope required to calculate MRT.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

95. Secondary Outcome: MRT for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

96. Secondary Outcome: MRT for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

97. Secondary Outcome: MRT for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

98. Secondary Outcome: MRT for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

99. Secondary Outcome: MRT for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

100. Secondary Outcome: MRT for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

101. Secondary Outcome: MRT for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 94
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

102. Secondary Outcome: Terminal Elimination Rate (Lambda z) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for lambda z as there were not enough data points collected for a terminal slope required to calculate lambda z.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

103. Secondary Outcome: Lambda z for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

104. Secondary Outcome: Lambda z for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

105. Secondary Outcome: Lambda z for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

106. Secondary Outcome: Lambda z for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

107. Secondary Outcome: Lambda z for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

108. Secondary Outcome: Lambda z for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

109. Secondary Outcome: Lambda z for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 102
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

110. Secondary Outcome: Terminal Phase Half-life (t1/2) for GSK2831781 0.0003 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12 and 24 hours post-dose
Population: PK population. Data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

111. Secondary Outcome: t1/2 for GSK2831781 0.0015 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

112. Secondary Outcome: t1/2 for GSK2831781 0.0075 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8 and 15 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

113. Secondary Outcome: t1/2 for GSK2831781 0.04 mg/kg (ADA-ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 15, 22, 29, 43 and 57 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 0

114. Secondary Outcome: t1/2 for GSK2831781 0.15 mg/kg (ADA-ve) and (ADA+ve)
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43 and 85 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 0 | 0

115. Secondary Outcome: t1/2 for GSK2831781 0.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 43, 85 and 121 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 0

116. Secondary Outcome: t1/2 for GSK2831781 1.5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 36, 43, 57, 85 and 121 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 0

117. Secondary Outcome: t1/2 for GSK2831781 5 mg/kg
Description: Blood samples were collected at specified time points for GSK2831781 in plasma.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours, Days 8, 11, 15, 18, 22, 29, 43, 57, 71, 85 and 121 post-dose
Population: as for outcome 110
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 0

118. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 in Healthy Volunteer Placebo
Description: Serum samples were collected at indicated time points for determination of ADA. ADAs to GSK2831781 was detected using a validated binding antibody detection.
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 191)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Healthy Volunteer Combined
Number analyzed (Participants) | 14
Participants
  Pre-dose | 3
  168 hours | 3
  Day 29 | 3
  Day 85 | 2
  Follow-up (Day 191) | 1

119. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.0003 mg/kg (ADA-ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, and follow-up (Day 29)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0003 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Participants
  Pre-dose | 0
  168 hours | 0
  Follow-up (Day 29) | 0

120. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.0015 mg/kg (ADA-ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29 and follow-up (Day 43)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0015 mg/kg (ADA-ve)
Number analyzed (Participants) | 1
Participants
  Pre-dose | 0
  168 hours | 0
  Day 29 | 0
  Follow-up (Day 43) | 0

121. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.0075 mg/kg (ADA-ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29 and follow-up (Day 85)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.0075 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Pre-dose | 1
  168 hours | 0
  Day 29 | 1
  Follow-up (Day 85) | 1

122. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.04 mg/kg (ADA-ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 147)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.04 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Pre-dose | 0
  168 hours | 0
  Day 29 | 1
  Day 85 | 0
  Follow-up (Day 147) | 0

123. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.15 mg/kg (ADA-ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 219)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.15 mg/kg (ADA-ve)
Number analyzed (Participants) | 6
Participants
  Pre-dose | 0
  168 hours | 2
  Day 29 | 1
  Day 85 | 1
  Follow-up (Day 219) | 0

124. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.15 mg/kg (ADA+ve)
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 191)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.15 mg/kg (ADA+ve)
Number analyzed (Participants) | 6
Participants
  Pre-dose | 6
  168 hours | 6
  Day 29 | 6
  Day 85 | 4
  Follow-up (Day 191) | 4

125. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 Placebo in Psoriasis Participants
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 307)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for Psoriasis
Number analyzed (Participants) | 9
Participants
  Pre-dose | 1
  168 hours | 1
  Day 29 | 1
  Day 85 | 1
  Follow-up (Day 307) | 1

126. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 0.5 mg/kg
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 237)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 0.5 mg/kg
Number analyzed (Participants) | 6
Participants
  Pre-dose | 0
  168 hours | 1
  Day 29 | 1
  Day 85 | 2
  Follow-up (Day 237) | 1

127. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 1.5 mg/kg
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 277)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 1.5 mg/kg
Number analyzed (Participants) | 6
Participants
  Pre-dose | 1
  168 hours | 1
  Day 29 | 1
  Day 85 | 1
  Follow-up (Day 277) | 1

128. Secondary Outcome: Number of Participants With Positive ADAs to GSK2831781 5 mg/kg
Description: as for outcome 118
Time Frame: Pre-dose (Day 1), 168 hours, Days 29, 85 and follow-up (Day 307)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2831781 5 mg/kg
Number analyzed (Participants) | 6
Participants
  Pre-dose | 0
  168 hours | 0
  Day 29 | 0
  Day 85 | 1
  Follow-up (Day 307) | 1

129. Secondary Outcome: Change From Baseline in Psoriasis Area Severity Index (PASI) Scores
Description: PASI score was determined by evaluation of body surface area (BSA) covered by plaque psoriasis in 4 areas (head, upper extremities, trunk and lower extremities with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged from 0=No symptoms, 1=slight, 2=moderate, 3=marked and 4=very marked) of erythema, induration and scaling in each of the 4 areas. PASI score ranges from 0 (no psoriasis) to 72 (worse psoriasis). Final PASI=(sum of severity score for each area) * (% body area affected score * area score). Baseline was considered as the latest pre-dose assessment with a non-missing value for Day -1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Day 15 (n=9,6,6,6) | -0.7 (2.66) | -1.7 (2.43) | -2.4 (2.56) | -2.7 (2.54)
  Day 29 (n=9,6,6,6) | -0.5 (3.09) | -1.8 (2.25) | -3.3 (4.53) | -3.5 (2.93)
  Day 43 (n=9,6,6,6) | -1.7 (4.12) | -1.6 (2.40) | -3.8 (4.36) | -3.7 (2.66)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | -1.0 (6.09) |  | 1.2 (3.75) | -3.3 (2.55)
  Day 121 (n=9,6,6,6) | -0.6 (3.03) | -0.5 (2.44) | 1.2 (5.83) | -2.7 (2.21)

130. Secondary Outcome: Actual PASI Scores
Description: PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head, upper extremities, trunk and lower extremities with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged from 0=No symptoms, 1=slight, 2=moderate, 3=marked and 4=very marked) of erythema, induration and scaling in each of the 4 areas. PASI score ranges from 0 (no psoriasis) to 72 (worse psoriasis). Final PASI=(sum of severity score for each area) * (% body area affected score * area score).
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Baseline (n=9,6,6,6) | 10.3 (4.52) | 6.8 (2.40) | 14.1 (6.55) | 9.2 (4.09)
  Day 15 (n=9,6,6,6) | 9.6 (3.92) | 5.1 (2.84) | 11.7 (5.67) | 6.5 (2.98)
  Day 29 (n=9,6,6,6) | 9.8 (4.17) | 5.0 (2.82) | 10.8 (4.14) | 5.7 (2.54)
  Day 43 (n=9,6,6,6) | 8.6 (3.79) | 5.2 (2.71) | 10.4 (4.06) | 5.5 (2.20)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | 9.4 (5.94) |  | 15.4 (6.73) | 5.9 (2.39)
  Day 121 (n=9,6,6,6) | 9.8 (5.20) | 6.3 (3.00) | 15.4 (8.59) | 6.5 (3.76)

131. Secondary Outcome: Percentage of Participants Who Achieved >=50 Percent (%) and >=75% Improvement From Baseline in PASI Score
Description: PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head, upper extremities, trunk and lower extremities with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged from 0=No symptoms, 1=slight, 2=moderate, 3=marked and 4=very marked) of erythema, induration and scaling in each of the 4 areas. PASI score ranges from 0 (no psoriasis) to 72 (worse psoriasis). Final PASI=(sum of severity score for each area) * (% body area affected score * area score). Baseline was considered as the latest pre-dose assessment with a non-missing value for Day -1.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Percentage of participants
  PASI 50: Day 15 (n=9,6,6,6) | 0 | 17 | 0 | 17
  PASI 50: Day 29 (n=9,6,6,6) | 0 | 33 | 17 | 17
  PASI 50: Day 43 (n=9,6,6,6) | 11 | 33 | 17 | 33
  PASI 50: Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  PASI 50: Day 85 (n=6,0,6,6) | 17 |  | 0 | 17
  PASI 50: Day 121 (n=9,6,6,6) | 11 | 17 | 0 | 0
  PASI 75: Day 15 (n=9,6,6,6) | 0 | 0 | 0 | 0
  PASI 75: Day 29 (n=9,6,6,6) | 0 | 0 | 0 | 0
  PASI 75: Day 43 (n=9,6,6,6) | 0 | 0 | 0 | 0
  PASI 75: Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  PASI 75: Day 85 (n=6,0,6,6) | 0 |  | 0 | 0
  PASI 75: Day 121 (n=9,6,6,6) | 0 | 17 | 0 | 0

132. Secondary Outcome: Change From Baseline in Plaque Lesional Severity Score (PLSS) Scores for the Index Plaque
Description: PLSS is a 0 to 12 point rating scale for lesions, calculated as the sum of the scores (ranging from 0 = no symptoms to 4 = very marked) for 3 symptoms: induration, erythema and scaling, measured by a qualified dermatologist. The PLSS score for the Index Plaque ranged from 0 to 12. The score 0 indicated no symptoms and 12 is the worst score. Baseline was considered as the latest pre-dose assessment with a non-missing value for Day -1. Change from Baseline was calculated as post-Baseline value minus Baseline value. A negative change from Baseline is an improvement in symptoms.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Day 15 (n=9,6,6,6) | -0.6 (1.24) | -1.3 (1.03) | -1.8 (1.47) | -1.7 (1.03)
  Day 29 (n=9,6,6,6) | -0.2 (1.79) | -2.2 (1.33) | -1.8 (1.47) | -2.0 (0.89)
  Day 43 (n=9,6,6,6) | -0.7 (2.00) | -1.8 (1.17) | -1.8 (1.47) | -1.8 (1.17)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | -1.7 (2.42) |  | -1.2 (2.04) | -1.5 (1.64)
  Day 121 (n=9,6,6,6) | -0.9 (2.42) | -0.5 (1.38) | -1.2 (2.64) | -0.7 (1.63)

133. Secondary Outcome: Absolute PLSS Scores for the Index Plaque
Description: PLSS is a 0 to 12 point rating scale for lesions, calculated as the sum of the scores (ranging from 0 = no symptoms to 4 = very marked) for 3 symptoms: induration, erythema and scaling, measured by a qualified dermatologist. The PLSS score for the Index Plaque ranged from 0 to 12. The score 0 indicated no symptoms and 12 is the worst score.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Baseline (n=9,6,6,6) | 7.1 (1.05) | 6.5 (1.38) | 7.7 (1.37) | 6.5 (0.84)
  Day 15 (n=9,6,6,6) | 6.6 (1.24) | 5.2 (1.94) | 5.8 (1.72) | 4.8 (1.33)
  Day 29 (n=9,6,6,6) | 6.9 (14.62) | 4.3 (1.75) | 5.8 (1.72) | 4.5 (1.05)
  Day 43 (n=9,6,6,6) | 6.4 (2.19) | 4.7 (1.97) | 5.8 (1.72) | 4.7 (1.21)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | 5.7 (3.39) |  | 6.5 (1.05) | 5.0 (1.67)
  Day 121 (n=9,6,6,6) | 6.2 (2.54) | 6.0 (1.41) | 6.5 (1.76) | 5.8 (1.17)

134. Secondary Outcome: Change From Baseline in Physicians Global Assessment (PGA) Scores in Psoriasis Participants
Description: A 7-point scoring system was used to measure the severity of psoriatic lesions over the whole body. The score 0 indicated as clear: no signs of psoriasis and 6 indicated as severe: very marked plaque elevation, scaling and erythema. Baseline was considered as the latest pre-dose assessment with a non-missing value for Day -1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Day 15 (n=9,6,6,6) | -0.1 (1.05) | -0.7 (0.82) | -0.3 (0.82) | -1.0 (0.63)
  Day 29 (n=9,6,6,6) | -0.3 (1.58) | -0.5 (0.84) | -0.5 (1.05) | -1.3 (1.03)
  Day 43 (n=9,6,6,6) | -0.4 (1.59) | 0.0 (0.89) | -0.8 (0.98) | -1.5 (0.55)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | -0.7 (2.07) |  | 0.0 (0.89) | -1.5 (0.55)
  Day 121 (n=9,6,6,6) | -0.3 (1.50) | 0.7 (1.75) | -0.3 (1.21) | -1.0 (0.00)

135. Secondary Outcome: Absolute PGA Scores in Psoriasis Participants
Description: A 7-point scoring system was used to measure the severity of psoriatic lesions over the whole body. The score 0 indicated as clear: no signs of psoriasis and 6 indicated as severe: very marked plaque elevation, scaling and erythema.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Scores on a scale
  Baseline (n=9,6,6,6) | 4.4 (0.88) | 3.2 (0.75) | 4.8 (0.75) | 4.2 (0.98)
  Day 15 (n=9,6,6,6) | 4.3 (0.71) | 2.5 (1.05) | 4.5 (1.05) | 3.2 (1.17)
  Day 29 (n=9,6,6,6) | 4.1 (1.05) | 2.7 (0.82) | 4.3 (1.21) | 2.8 (0.75)
  Day 43 (n=9,6,6,6) | 4.0 (1.12) | 3.2 (0.75) | 4.0 (0.89) | 2.7 (0.52)
  Day 85 (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day 85 (n=6,0,6,6) | 4.0 (1.79) |  | 4.8 (0.98) | 2.7 (0.52)
  Day 121 (n=9,6,6,6) | 4.1 (1.36) | 3.8 (1.47) | 4.5 (1.38) | 3.2 (0.98)

136. Secondary Outcome: Percentage of Participants in Each PGA Score Category
Description: A 7-point scoring system was used to measure the severity of psoriatic lesions over the whole body. The score 0=clear, 1=almost clear, 2=mild, 3=mild to moderate, 4=moderate, 5=moderate to severe and 6=severe.
Time Frame: Baseline, Days 15, 29, 43, 85 and 121
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
Number analyzed (Participants) | 9 | 6 | 6 | 6
Percentage of participants
  Baseline:Almost clear(n=9,6,6,6) | 0 | 0 | 0 | 0
  Baseline:Mild (n=9,6,6,6) | 0 | 17 | 0 | 0
  Baseline:Mild to moderate(n=9,6,6,6) | 11 | 50 | 0 | 33
  Baseline:Moderate (n=9,6,6,6) | 44 | 33 | 33 | 17
  Baseline:Moderate to sever(n=9,6,6,6) | 33 | 0 | 50 | 50
  Baseline:Severe (n=9,6,6,6) | 11 | 0 | 17 | 0
  Day15:Almost clear(n=9,6,6,6) | 0 | 17 | 0 | 0
  Day15:Mild (n=9,6,6,6) | 0 | 33 | 0 | 33
  Day15:Mild to moderate(n=9,6,6,6) | 11 | 33 | 17 | 33
  Day15:Moderate (n=9,6,6,6) | 44 | 17 | 33 | 17
  Day15:Moderate to severe(n=9,6,6,6) | 44 | 0 | 33 | 17
  Day15:Severe (n=9,6,6,6) | 0 | 0 | 17 | 0
  Day29:Almost clear(n=9,6,6,6) | 0 | 0 | 0 | 0
  Day29:Mild (n=9,6,6,6) | 0 | 50 | 0 | 33
  Day29:Mild to moderate(n=9,6,6,6) | 33 | 33 | 33 | 50
  Day29:Moderate (n=9,6,6,6) | 33 | 17 | 17 | 17
  Day29:Moderate to severe(n=9,6,6,6) | 22 | 0 | 33 | 0
  Day29:Severe (n=9,6,6,6) | 11 | 0 | 17 | 0
  Day43:Almost clear(n=9,6,6,6) | 0 | 0 | 0 | 0
  Day43:Mild (n=9,6,6,6) | 0 | 17 | 0 | 33
  Day43:Mild to moderate(n=9,6,6,6) | 44 | 50 | 33 | 67
  Day43:Moderate (n=9,6,6,6) | 22 | 33 | 33 | 0
  Day43:Moderate to severe(n=9,6,6,6) | 22 | 0 | 33 | 0
  Day43:Severe (n=9,6,6,6) | 11 | 0 | 0 | 0
  Day85:Almost clear(n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Almost clear(n=6,0,6,6) | 17 |  | 0 | 0
  Day85:Mild (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Mild (n=6,0,6,6) | 0 |  | 0 | 33
  Day85:Mild to moderate(n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Mild to moderate(n=6,0,6,6) | 17 |  | 0 | 67
  Day85:Moderate (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Moderate (n=6,0,6,6) | 17 |  | 50 | 0
  Day85:Moderate to severe(n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Moderate to severe(n=6,0,6,6) | 33 |  | 17 | 0
  Day85:Severe (n=6,0,6,6): number analyzed (Participants) | 6 | 0 | 6 | 6
  Day85:Severe (n=6,0,6,6) | 17 |  | 33 | 0
  Day121:Almost clear(n=9,6,6,6) | 11 | 17 | 0 | 0
  Day121:Mild (n=9,6,6,6) | 0 | 0 | 0 | 33
  Day121:Mild to moderate(n=9,6,6,6) | 11 | 0 | 33 | 17
  Day121:Moderate (n=9,6,6,6) | 22 | 50 | 17 | 50
  Day121:Moderate to severe(n=9,6,6,6) | 56 | 33 | 17 | 0
  Day121:Severe (n=9,6,6,6) | 0 | 0 | 33 | 0

ADVERSE EVENTS:
Time Frame: On treatment AEs and SAEs were collected Up to 307 days
Description: Safety population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo for Healthy Volunteer Combined | GSK2831781 0.0003 mg/kg (ADA-ve) | GSK2831781 0.0015 mg/kg (ADA-ve) | GSK2831781 0.0075 mg/kg (ADA-ve) | GSK2831781 0.04 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA-ve) | GSK2831781 0.15 mg/kg (ADA+ve) | Placebo for Psoriasis | GSK2831781 0.5 mg/kg | GSK2831781 1.5 mg/kg | GSK2831781 5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 8/14 | 0/1 | 0/1 | 5/6 | 6/6 | 3/6 | 3/6 | 9/9 | 4/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for Healthy Volunteer Combined (N=14) | GSK2831781 0.0003 mg/kg (ADA-ve) (N=1) | GSK2831781 0.0015 mg/kg (ADA-ve) (N=1) | GSK2831781 0.0075 mg/kg (ADA-ve) (N=6) | GSK2831781 0.04 mg/kg (ADA-ve) (N=6) | GSK2831781 0.15 mg/kg (ADA-ve) (N=6) | GSK2831781 0.15 mg/kg (ADA+ve) (N=6) | Placebo for Psoriasis (N=9) | GSK2831781 0.5 mg/kg (N=6) | GSK2831781 1.5 mg/kg (N=6) | GSK2831781 5 mg/kg (N=6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for Healthy Volunteer Combined (N=14) | GSK2831781 0.0003 mg/kg (ADA-ve) (N=1) | GSK2831781 0.0015 mg/kg (ADA-ve) (N=1) | GSK2831781 0.0075 mg/kg (ADA-ve) (N=6) | GSK2831781 0.04 mg/kg (ADA-ve) (N=6) | GSK2831781 0.15 mg/kg (ADA-ve) (N=6) | GSK2831781 0.15 mg/kg (ADA+ve) (N=6) | Placebo for Psoriasis (N=9) | GSK2831781 0.5 mg/kg (N=6) | GSK2831781 1.5 mg/kg (N=6) | GSK2831781 5 mg/kg (N=6)
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 2 | 2 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 4 | 1 | 3 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Reticulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental care (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02195349/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02195349/SAP_001.pdf